CLINICAL TRIAL: NCT05290727
Title: Evaluation of the Efficacy of "Aquoral Lipo" Artificial Tears in Contact Lens Wearers With Discomfort Symptoms
Brief Title: Efficacy of "Aquoral Lipo" Artificial Tears in Contact Lens Wearers With Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Collaborators: Esteve (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IOBA-2021-54
Record Dates: First submitted 2022-02-22; First posted 2022-03-22 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Contact Lens Complication
Keywords: Contact lens; Discomfort; Artificial tears
MeSH Terms: interventions — hylan; Liposomes; crocin; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Low intervention level, prospective, crossover, double masked, randomized, single center clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study and control products will lack any identification label, except that concerning the assignment code. The product together with the instillation instructions will be delivered in a sealed envelope which will contain an identification label of the assignment code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.15% Aquoral Lipo (Esteve) and 0.15% Hyabak (Thea) (Other): Dosage form: topical administration multidose ophthalmic eye drops Product usage order will be determined through randomization Duration: 15 days + 15 days Frequency: dosage between 3 and 6 drops per day
  Interventions: Other: Aquoral Lipo (Esteve); Other: Hyabak (Thea)
- 0.15% Hyabak (Thea) and 0.15% Aquoral Lipo (Esteve) (Other): Dosage form: topical administration multidose ophthalmic eye drops Product usage order will be determined through randomization Duration: 15 days + 15 days Frequency: dosage between 3 and 6 drops per day
  Interventions: Other: Aquoral Lipo (Esteve); Other: Hyabak (Thea)

INTERVENTIONS:
Other: Aquoral Lipo (Esteve) — 15-day randomized treatment period of each of the clinical trial products (experimental and control) with a 1-week washout period prior to use of the study products
  Other Names: 0.15% Hyaluronic Acid crosslinked with liposomes and crocin
Other: Hyabak (Thea) — 15-day randomized treatment period of each of the clinical trial products (experimental and control) with a 1-week washout period prior to use of the study products
  Other Names: 0.15% Hyaluronic Acid

SUMMARY:
There are more than 140 million contact lens wearers in the world. However, contact lens use can cause discomfort symptoms in up to 50% of wearers. And these symptoms can lead to contact lens abandonment in 12-51% of symptomatic wearers.

Contact lens discomfort is defined by the Tear Film & Ocular Surface Society (TFOS) as a condition characterized by episodic or persistent adverse ocular sensations related to contact lens wear, either with or without visual disturbance, resulting from reduced compatibility between the contact lens and the ocular environment, which can lead to decreased wearing time and discontinuation of contact lens wear.

The most common cause of contact lens discontinuation is discomfort and dryness symptoms. This symptomatology is associated with visual acuity alterations, increased risk of ocular surface desiccation, or decreased contact lens wearing time. But the different signs found in contact lens wearers who present discomfort with contact lenses do not always correlate with the symptoms they report. In addition, different factors negatively impact contact lens discomfort such as low relative humidity environments.

In order to alleviate contact lens discomfort, the first option chosen by professionals is fitting another contact lens with different replacement frequency or material. The second option is recommending the use of lubricants or moisturizers, and the third one is changing the maintenance system.

The use of artificial tears is an effective way to improve contact lens discomfort, mainly by instilling them prior to contact lens insertion, since it provides the moisturizing factor that maintenance solutions lack. In addition, it improves comfort, visual quality, and reduces the production of deposits on the contact lens.

The hypothesis of this clinical trial is that "Aquoral Lipo" artificial tears are more effective than control artificial tears to improve symptomatology in contact lens wearers with discomfort symptoms.

The study will compare the effect of both "Aquoral Lipo" and control artificial tears under controlled normal and adverse environmental conditions.

DETAILED DESCRIPTION:
Justification:

The number of contact lens wearers is increasing every year. It is estimated that there are approximately more than 140 million wearers worldwide. However, around 50% of them suffer from discomfort while wearing their lenses, and 12-51% of them stop wearing contact lenses. The most common experienced symptoms are dry eye, redness, foreign body sensation, poor vision, or sensitivity to light.

Contact lens discomfort is defined by the Tear Film & Ocular Surface Society (TFOS) as a condition characterized by episodic or persistent adverse ocular sensations related to contact lens wear, either with or without visual disturbance, resulting from reduced compatibility between the contact lens and the ocular environment, which can lead to decreased wearing time and discontinuation of contact lens wear.

Symptoms related to contact lens discomfort can be associated with visual acuity alterations, increased risk of ocular surface desiccation, or decreased contact lens wearing time. But the majority of subjects who develop discomfort with contact lenses do not have associated ocular pathology or damage.

Contact lens discomfort can be caused by factors associated with the contact lens itself, such as material, design, and maintenance systems; and factors associated with the environment surrounding the contact lens, such as those of the wearer or environmental conditions.

In order to alleviate contact lens discomfort, 47% of professionals refit another contact lens of a different material or replacement frequency. 22% of professionals recommend the use of lubricants or moisturizers, and 15% change the maintenance system.

The use of artificial tears improves contact lens discomfort, mainly by instilling them prior to contact lens insertion, since it provides the moisturizing factor that maintenance solutions lack. During contact lens wear, they also improve comfort, visual quality, and reduce the production of contact lens deposits.

Aquoral Lipo is a preservative-free lubricant and antioxidant ophthalmic solution based on sodium salt of cross-linked hyaluronic acid, liposomes, and crocin. It provides good hydration and a long permanence time on the ocular surface.

Hypothesis:

"Aquoral Lipo" artificial tears are more effective than control artificial tears to improve symptomatology in contact lens wearers that suffer from discomfort symptoms.

Objective:

To compare the efficacy of Aquoral Lipo artificial tears with a product with 0.15% hyaluronic acid after 15 days of use in subjects with contact lens discomfort, and exposed to normal and adverse controlled conditions created in a controlled environment chamber.

Study plan:

Participants will perform a total of 5 visits (in 5 days): an inclusion visit (V0), two basal visits (V1 and V3), and two study visits (V2 and V4).

V0: Recruitment visit. Contact lens wearers will be recruited after checking inclusion and exclusion criteria. If eligible, participants will sign the informed consent and will be scheduled for V1 within the next 7 days.

V1: Baseline visit. Participants will come to the visit with a new pair of contact lenses and having worn them for at least 2 hours. Participants will enter the environmental chamber at the Controlled Environment Laboratory (CELab), where they will be exposed for 30 minutes to a normal controlled environment (23 degrees Celsius and 50 percentage relative humidity). Then, tests will be performed, and one of the study products will be dispensed to the subject randomly to be instilled 3-6 times a day until the next visit. Participants will come to the next visit within 15 days.

V2: Study visit (V2 NE - V2 AE). Participants will come to the visit having worn the contact lenses the same number of hours as in V1, and they will be exposed for 30 minutes to a normal controlled environment at CELab (V2 NE). Then, tests will be performed, and they will be exposed for 90 minutes to an adverse controlled environment (23 degrees Celsius and 10 percentage relative humidity) at CELab (V2 AE). Test will be repeated at 30, 60, and 90 minutes of the adverse environmental exposure. Subjects will not use artificial tears until the next visit, within the next 7 days.

V3: Baseline visit. The same procedures as in V1 will be followed, but the other study product will be dispensed to participants to be instilled 3-6 times a day until the next visit, within 15 days.

V4: Study visit (V4 NE - V4 AE). The same procedures as in V2 will be followed.

Clinical evaluation:

* Contact lens discomfort symptoms questionnaires
* Visual Acuity measurement
* Tear film lipid layer thickness measurement (interferometry)
* Blinking measurement
* Evaporimetry
* Non Invasive Break Up Time (NIBUT)
* Anterior pole biomicroscopy
* Tear Break Up Time with fluorescein (TBUT)
* Corneal staining with fluorescein
* Conjunctival staining with lissamine green

Data analysis:

Means and standard deviations will be calculated for the quantitative variables of the study. For ordinal variables, medians and interquartile ranges will be calculated. Qualitative variables will be summarized using percentages together with their confidence intervals.

For primary efficacy endpoint, CLDEQ-8 comparisons between V1 and V2 NE, and V3 and V4 NE will be performed by t-Student test for two paired samples.

The evolution of all variables over time will be analyzed through an ANOVA for repeated measures. Their evolution after the exposure to adverse environments will be analyzed through Student's t-test for paired samples (quantitative variables) and McNemar's test (ordinal variables).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Signature of informed consent form
* Regular hydrophilic contact lens wearers: at least 4 times a week and at least 4 hours a day
* Contact lens discomfort measured as a Contact Lens Dry Eye Questionnaire-8 score higher than 11 points

Exclusion Criteria:

* Known sensitivity or intolerance to some of the products used in the study
* Habitual non-compliance of the contact lens replacement frequency
* Any systemic disease or treatment that alters the eye
* Any ocular surgery, infection, inflammation, or active eye disease, in the last year
* Autoimmune dry eye
* Participation in a clinical trial within 30 days prior to entry into this study
* Pregnancy or breastfeeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
The Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) | After the use of the study product (15 days from treatment start)
  Significant changes of at least 3 points in the questionnaire between the two products (study and control).
  This questionnaire quantifies the symptoms of ocular discomfort during the use of contact lenses. Values up to 37 points are obtained, with higher values representing greater symptomatology.

SECONDARY OUTCOMES:
The CLDEQ-8 | After the use of the study product (15 days from treatment start)
  Significant changes after exposure to normal and adverse environments. This questionnaire quantifies the symptoms of ocular discomfort during the use of contact lenses. Values up to 37 points are obtained, with higher values representing greater symptomatology.
The Contact Lens Discomfort Index | After the use of the study product (15 days from treatment start)
  Significant changes after exposure to normal and adverse environments. This questionnaire allows establishing the presence of contact lens discomfort according to its symptoms. Values up to 18 points are obtained, with higher values representing greater symptomatology.
Comfort and dryness Visual Assessment Scales | After the use of the study product (15 days from treatment start)
  Significant changes after exposure to normal and adverse environments. Visual Assessment Scales evaluate ocular comfort and dryness during contact lens wear by using a horizontal straight line of 100 mm that allows assessment on a scale of 0 to 100 points (higher values indicating greater symptoms).
Tear film stability | After the use of the study product (15 days from treatment start)
  Significant changes after exposure to normal and adverse environments. Tear break up time will be evaluated by instilling fluorescein sodium in the inferior conjunctival fornix. Tear film pattern will be observed through a slit lamp with the cobalt blue filter, and through a #12 Wratten yellow filter. The time between the last blink and the moment when the first black spot appears will be noted in seconds.
Tear film evaporimetry | After the use of the study product (15 days from treatment start)
  Significant changes after exposure to normal and adverse environments. Tear evaporation rate (g/m²h) will be evaluated using a closed chamber evaporimeter without ventilation, the Eye Vapometer. The subject will be asked to blink normally and remain in the primary gaze position while measurements are taken with the eyes open and closed.
Tear film interferometry | After the use of the study product (15 days from treatment start)
  Significant changes after exposure to normal and adverse environments. The value of the lipid layer thickness obtained through the interferometric pattern of the tear film will be observed and measured in a scale of 0-100 nm.
Number of blinks | After the use of the study product (15 days from treatment start)
  Significant changes after exposure to normal and adverse environments. Number of times the subject blinks during a period of 20 seconds will be counted.
Corneal staining | After the use of the study product (15 days from treatment start)
  Significant changes in corneal staining after adverse environments. To assess corneal staining, fluorescein sodium will be instilled in the inferior conjunctival fornix. The surface of the cornea will be examined under a slit lamp through the cobalt blue and a #12 Wratten yellow filters. The intensity of the corneal fluorescein staining will be graded on a scale of 0 to 4 degrees according to the Oxford scale.
Conjunctival staining | After the use of the study product (15 days from treatment start)
  Significant changes in conjunctival staining after adverse environments. Lissamine green strips will be used and moistened with physiological serum. They will be instilled by impregnating the superior bulbar conjunctiva. Nasal and temporal conjunctival areas will be evaluated and assessed on a scale of 0 to 4 degrees according to the Oxford scale.
Hours of contact lens wear | After the use of the study product (15 days from treatment start)
  Significant changes in the time of contact lens wear will be evaluated.
Comfortable hours of contact lens wear | After the use of the study product (15 days from treatment start)
  Significant changes in the number of hours the patient is comfortable with contact lens wear.
Number of daily instillations of the products | After the use of the study product (15 days from treatment start)
  Significant changes in the number of daily products instillations.
User satisfaction with the products | After the use of the study product (15 days from treatment start)
  Significant changes in the products satisfaction. Satisfaction with the products will be assessed on a horizontal line of 100 mm and graded between 0-10 points. The left end indicates the subject is extremely dissatisfied and the right end indicates the subject is extremely satisfied. The evaluation will be carried out by measuring with a millimeter ruler the distance from the left end, giving it a value of "zero", to the right with a value of "one hundred".

OTHER OUTCOMES:
Visual acuity | 45 days after screening visit
  Changes of at least one line of visual acuity not improvable with correction or instillation of artificial tears.
  Visual acuity will be measured monocularly using the Age-Related Eye Disease Study (AREDS) Study Group modification of the Diabetic Retinopathy Early Treatment Study Group (ETDRS) method, at a distance of 4 meters.
Presence of ocular or periorbital adverse events | 45 days after screening visit
  The frequency of adverse events between the two study products (experimental and control) and the percentage of events that involves the withdrawal of patients from the study will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- IOBA - University of Valladolid, Valladolid, Spain